CLINICAL TRIAL: NCT04432740
Title: Clinical Outcomes Comparison of Distal Radius Fractures Between Two Conservative Treatment Methods: Below-Arm Cast Versus Reverse Sugar Tong Splint
Brief Title: A Novel Splint Technique for Distal Radius Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Çamur, Principal Investigator, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/45
Record Dates: First submitted 2020-05-29; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Distal Radius Fracture; Complication of Treatment
Keywords: distal radius fracture; conservative treatment; reverse sugar tong; below arm cast
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Below Arm Cast Group (Active Comparator): All the patients were prepared in the supine position at the emergency department. For analgesia, we used the hematoma block technique with 3 cc of 2% prilocaine hydrochloride®. In this group, after traction was applied using a finger-trap traction with a 4.5 kg weight for 5 minutes, the standard below arm cast was applied. Patients were encouraged to actively move their fingers, ipsilateral shoulder, and elbow in all the groups. Both treatments lasted 5 or 6 weeks after at our clinic
  Interventions: Procedure: Conservative Treatment of Distal Radius Fracture
- Reverse Sugar Tong Group (Active Comparator): In this group, after traction was applied using a finger-trap traction with a 4.5 kg weight for 5 minutes, sugar tong splint made of 12 layers of plaster was performed by one person. The reverse sugar tong splint succeeds as a classic sugar tong splint by stabilizing the volar and dorsal aspects of the wrist and forearm, maintaining the same degree of immobilization. The splint fold is located distally at the first web space of the hand, which does not immobilize the elbow. In all the groups, the wrist immobilization position was the same; pronated forearm, 15-20° wrist flexion, ulnar deviation, and care was taken not to immobilize the metacarpophalangeal joints. Patients were encouraged to actively move their fingers, ipsilateral shoulder, and elbow in all the groups. Both treatments lasted 5 or 6 weeks after at our clinic
  Interventions: Procedure: Conservative Treatment of Distal Radius Fracture

INTERVENTIONS:
Procedure: Conservative Treatment of Distal Radius Fracture — The purpose of this prospective randomized study was to compare a new reverse sugar tong splint technique that does not immobilize the elbow with a below-arm cast, in terms of patient radiological and clinical outcomes and the ability to maintain fracture reduction.

SUMMARY:
There are many conservative treatment methods, including below arm cast, above arm cast, and sugar tong splint that aim to obtain maximum functional, clinical, and radiological results There are no clear indications with regard to the best treatment including conservative or surgical methods for the different fracture subtypes in distal radius fracture. The purpose of this prospective randomized study was to compare a new reverse sugar tong splint technique that does not immobilize the elbow with a below-arm cast, in terms of patient radiological and clinical outcomes and the ability to maintain fracture reduction.

DETAILED DESCRIPTION:
This study was conducted at a single Orthopedics and Traumatology emergency department center between April 2017 and March 2019. A two-arm, parallel-group, prospective randomized trial was conducted to compare below-arm cast (BAC) and reverse sugar tong (RST) (described below) treatment of DRF.

Overall, 231 patients diagnosed with distal radius fracture in the emergency department received prospective treatment.

Inclusion criteria: Patients aged >18 years and with distal radius fracture type A and B (who presented within 10 days of the injury) were considered for inclusion.

Exclusion criteria: Patients with AO type C distal radius fractures (treated surgically), type 2 and 3 open fractures (according to Gustilo classification), previous hand or wrist surgery, fractures in the concomitant side of the upper extremities, associate carpal fracture, deformity on same extremity, pathological fractures, and cognitive deficit that does not allow the patient to understand the functional evaluation were excluded from this study. Lastly, patients who did not return for a follow-up visit at the end of the cast or splint treatment were also excluded.

Patient selection and treatment methods Sample Size: The sample size was calculated based on a 15-20% difference in complication rate between the two treatment groups, an alpha level of 5% and a power of 80%. Consequently, each group shall at least consist of 55 participants. We considered an extra 20% who loss of follow-up or loss of reduction and surgery may require for balancing sample size. With expectation of dropouts70 patients per group were included.

All the initial fractures of the patients were classified by the same author using the AO classification. Patients were randomly allocated to a treatment group using an electronic random number generator, with those having an even number assigned to the BAC group and those having an odd number to the RST group. Treatment in both the BAC and RST groups was conducted by the same investigator. The reduction obtained was checked on AP and lateral x-ray of the wrist, which were then used to calculate the following baseline radiological parameters: radial inclination (RI), radial height (RH), and volar tilt (VT).

Follow-up Management Clinical and radiological follow-up was performed 7-10 days (initial follow-up), three weeks, 5 or 6 weeks, 12 weeks and one year (last follow-up) after the treatment. X-rays at the initial follow-up which was performed 7-10 days after the initial closed reduction were taken with the cast or splint in place. Maintenance of fracture reduction was defined as a loss of reduction of less than 2 mm of radial height, 5° of radial inclination or 10° of volar tilt from the initial reduction films, and/or less than 2 mm of intra-articular step-off. In the initial follow-up, third week, and 6th week visit, patients were evaluated with x-ray to detect cast and splint complications, including those that require cast wedging or valving to reduce the pressure and the presence of complex regional pain syndrome (CRPS). Both treatments were removed during the 5-6th week visit in all groups.

Functional outcomes The validated quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) questionnaire score and the Mayo Elbow Performance score (MEPS) score were used to measure clinical outcomes.These scores were performed at the12th week and last follow-up visit for all the patients. Both groups were also evaluated with the Health Assessment Questionnaire (HAQ) at the 6th week visit for health status.

Radiological evaluation All the radiological parameters were measured by the same author at two time points: initial visit postreduction and 6th visit after the end of treatment. Radial height, Radial inclination and Volar tilt were measured separetly.

Clinical evaluations The wrist range of motion was measured in degree, using a goniometer, from the neutral position to flexion, extension, radial deviation, and ulnar deviation by same investigator during the last follow-up visit. The forearm rotation was also measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years,
* with distal radius fracture type A and B (who presented within 10 days of the injury)

Exclusion Criteria:

* Patients with AO type C distal radius fractures (treated surgically),
* type 2 and 3 open fractures (according to Gustilo classification),
* previous hand or wrist surgery,
* fractures in the concomitant side of the upper extremities,
* associate carpal fracture, deformity on the same extremity,
* pathological fractures,
* cognitive deficit that does not allow the patient to understand the functional evaluation
* patients who did not return for a follow-up visit at the end of the cast or splint treatment

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Fracture Healing Outcome | 6th week
  All patients were evaluated fracture healing with x-ray view which assessment of radiological union by observing the presence of bridging callus or the obscuration of the fracture line.

SECONDARY OUTCOMES:
Health relaated quality of life | 6th week
  Both groups were also evaluated with the Health Assessment Questionnaire (HAQ) for quality of life. The HAQ score is a feasible scale consisting of 8 different categories totally with 20 items which beneficial for assessing the functional disabilities during activities of daily living which is the increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment.
Rate of Complications Outcomes | 1st week, 3rd week and 6th week
  All patients were evaluated with x-ray to detect cast and splint complications, including those that loss of reduction, require cast wedging or valving to reduce the pressure and the presence of complex regional pain syndrome.
Functional Outcomes | 12th week and 1st year
  Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) questionnaire score was used to measure clinical outcomes.To calculate a QuickDASH score, at least 10 of the 11 items must be completed. Similar to the DASH, each item has 5 response options and, from the item scores, scale scores are calculated, ranging from 0 (no disability) to 100 (most severe disability).
Functional Outcomes | 12th week and 1st year
  Mayo Elbow Performance score (MEPS) score was used to measure clinical outcomes.The MEPS measures elbow function across four domains: pain (45 points), stability (10 points), range of motion (20 points), and daily functional tasks (25 points). Scores are categorized as 90-100 = excellent, 75-89 = good, 60-74 = fair, 0-59 = poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No